CLINICAL TRIAL: NCT04287114
Title: Cardiac Stroke Volume at Rest and During Different Exercise Intensities
Acronym: SVproject
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: T24/2020
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Function
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy young men and women (Experimental): Single group consisting of 10 men and 10 women
  Interventions: Behavioral: Acute exercise

INTERVENTIONS:
Behavioral: Acute exercise — Acute exercise with different exercise intensities

SUMMARY:
The main aim of the present investigation is to study cardiac function in different exercise intensities in healthy human subjects. Two techniques will be used: cardiac ultrasound-derived stroke volume measurements and body impedance measurements. 20 healthy men (n=10) and women (n=10) aged 18-45 years will be investigated at rest and during exercise. All study procedures are non-invasive.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* BMI 18-30
* Resting Blood pressure < 140/90 mmHg
* Participation in regular exercise

Exclusion Criteria:

* Acute illness
* Pregnancy
* Pace maker
* Artificial joint
* History of a cardiac event
* Insulin or medically treated diabetes
* Any chronic disease or condition that could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results
* Abundant use of alcohol
* Use of narcotics
* Smoking of tobacco or consuming snuff tobacco
* Diagnosed depressive or bipolar disorder
* Abnormalities in resting ECG (revised by the study physician)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac stroke volume | 1 min

SECONDARY OUTCOMES:
End-diastolic and end-systolic volumes | 1 min
Ejection fraction | 1 min

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Turku PET Centre, Turku
  - University of Turku, Turku

IPD SHARING:
Plan to Share IPD: No